CLINICAL TRIAL: NCT01897155
Title: Effect of Acute Arterial Hypertension on Morphine's Requirements and Postsurgical Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RIH_AP-UC-2012
Record Dates: First submitted 2013-01-19; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-06

CONDITIONS: Hypertensive Disease; Pain, Postoperative
Keywords: analgesia, postoperative;; analgesics opioid;; hyperalgesia;; remifentanil;; hypertension.
MeSH Terms: conditions — Hypertension; Pain, Postoperative; Agnosia; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBP 20-30% under baseline (Other): Induction of anesthesia was performed with remifentanil, pentothal 3 mg/kg and atracurium 0.5 mg/Kg. Anaesthesia was maintained with remifentanil (0.4 ug/Kg/min) and isoflurane adjusted to bispectral index (40-60). Patients received a phenylephrine infusion to maintain systolic blood pressure (SBP) 20% to 30% under baseline. The lower limit of SBP was 75 mmHg. In the recovery room, morphine was administered routinely at doses of 3 mg IV every 15 minutes until pain was less than 4 estimated by visual analog scale (VAS). VAS and pain threshold with von Frey filaments were assessed at 2, 6, 12 and 24 postoperative hours. All patients, received ketorolac 30 mg IV every 8 hours and intravenous morphine administered by patient controlled analgesia system (PCA) during the first 24 hours.
  Interventions: Other: SBP 20-30% over baseline
- SBP 20-30% over baseline (Other): Induction of anesthesia was performed with remifentanil, pentothal 3 mg/kg and atracurium 0.5 mg/Kg. Anaesthesia was maintained with remifentanil (0.4 ug/Kg/min) and isoflurane adjusted to bispectral index(40-60). Patients received a phenylephrine infusion in order to maintain systolic blood pressure (SBP) 20% to 30% over baseline. The upper limit of SBP was 165 mmHg. In the recovery room, morphine was administered routinely at doses of 3 mg IV every 15 minutes until pain was less than 4 estimated by visual analog scale (VAS). VAS and pain threshold with von Frey filaments were assessed at 2, 6, 12 and 24 postoperative hours. All patients, received ketorolac 30 mg IV every 8 hours and intravenous morphine administered by patient controlled analgesia system (PCA) during the first 24 hours.
  Interventions: Other: SBP 20-30% under baseline

INTERVENTIONS:
Other: SBP 20-30% over baseline — Patients were assigned to receive a phenylephrine infusion in order to maintain systolic blood pressure (SBP) 20% to 30% over the baseline. The upper limit of systolic blood pressure is 165 mmHg.
  Arms: SBP 20-30% under baseline
Other: SBP 20-30% under baseline — Patients were assigned to receive a phenylephrine infusion in order to maintain systolic blood pressure (SBP) 20% to 30% below the baseline. The lower limit of systolic blood pressure is 75 mmHg
  Arms: SBP 20-30% over baseline

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the effect of acute arterial hypertension maintained during surgery on morphine's requirements in patients undergoing laparoscopic cholecystectomy

DETAILED DESCRIPTION:
The high arterial blood pressure has been correlated with an increase in pain threshold in animal and humans. One of the explanations to this phenomenon is a baroreceptor activity and vasopressin release at the level of spinal cord dorsal horn and hypothalamus.

As far as we know, there is only one study about the effect of chronic hypertension on postoperative pain and none with acute hypertension. We therefore decided to conduct a randomized controlled trial to evaluate the effect of acute hypertension on postoperative morphine's requirements.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology patient classification status(ASA) I-II
* Between 20 and 60 years of age
* Programed for elective laparoscopic cholecystectomy

Exclusion Criteria:

* History of arterial hypertension
* Baseline blood pressure over 139/89
* Use of opioids and any analgesic drug during the last 24 hours before surgery
* Chronic use of nonsteroidal antiinflammatory
* BMI > 34.9
* History of drug or alcohol abuse
* Use of medications that interfere in the central nervous system
* Adverse reactions to the drugs used in the study
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Morphine requirement post laparoscopic cholecystectomy | First 24 hours postoperative
  Measure of morphine consumption during the first 24 postoperative hours in patients undergoing laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Effects of acute hypertension in pain scores | First 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Delfino, MD, Principal Investigator — Departamento de Anestesiología, Hospital Clínico Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica, Santiago, Santiago Metropolitan, Chile